CLINICAL TRIAL: NCT03284996
Title: Role of Doppler Ultrasound in Early Detection of Diabetic Nephropathy in Patients With Type 2 Diabetes Mellitus.
Brief Title: Doppler Ultrasound in Early Detection of Diabetic Nephropathy Type 2 Diabetes Mellitus.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shery Dawood Yassa, Principal investigator, Assiut University
Other Study IDs: DUDN
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Doppler ultrasonography — Examination of the whole cases & controls by doppler ultrasound to measure renal resistive index.

SUMMARY:
Doppler sonography provides an easily applicable, non-invasive, and well-established method for investigating renal morphologic characteristics and measuring vascular resistance in the renal parenchyma. Doppler are of strategic importance in providing qualitative and quantitative information about the renal vasculature, which can be obtained through the assessment of the resistive index.

DETAILED DESCRIPTION:
Nephropathy is one of the most common long-term, life-threatening complications causing a high rate of morbidity and mortality among individual patients with type 2 diabetes.

The onset and progression of nephropathy can be delayed by interventions, provided they are instituted early in the course of the disease.

Doppler sonography allows non-invasive method for investigating renal hemodynamics. Renal resistive index measured using Doppler ultrasonography, reflects intra-renal vascular resistance.

Although Doppler sonography clearly does not substitute for renal biopsy, several studies have suggested that it might aid in the management of established renal disease and provide an easily applicable and noninvasive method for investigating renal hemodynamics.

Doppler sonography provides an easily applicable, non-invasive, and well-established method for investigating renal morphologic characteristics and measuring vascular resistance in the renal parenchyma. Doppler are of strategic importance in providing qualitative and quantitative information about the renal vasculature, which can be obtained through the assessment of the resistive index. It is one of the most sensitive parameters in the study of kidney diseases and allows us to quantify the changes in renal plasma flow . A normal resistive index is below 0.7 in adults and children who are six years of age or older.

ELIGIBILITY:
Inclusion Criteria:

* 1. Type 2 diabetic patients. 2. Serum creatinine <1.2 mg/dl

Exclusion Criteria:

- 1. patients with known history of renal disease or any systemic diseases with renal complications.

2. Serum creatinine >1.2 mg/dl

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was designed as a single-center case control study in which we'll evaluate intra-renal hemodynamic changes with Doppler sonography in diabetic patients in comparison to non-diabetic controls, by studying 80 cases, 40 cases of patients with type 2 diabetes mellitus from the diabetes & nephrology outpatient clinic in Assiut University Hospital (group A) and 40 age-matched healthy adults served as a control group (group B).
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Early detection of diabetic nephropathy in patients with type 2 diabetes mellitus by measuring changes in renal resistive index using Doppler ultrasonography | 2 years
  Early detection of diabetic nephropathy in patients with type 2 diabetes mellitus by measuring changes in renal resistive index using Doppler ultrasonography

REFERENCES:
- [Result] Nelson TR, Pretorius DH. The Doppler signal: where does it come from and what does it mean? AJR Am J Roentgenol. 1988 Sep;151(3):439-47. doi: 10.2214/ajr.151.3.439. PMID 2970215
- [Result] Tublin ME, Bude RO, Platt JF. Review. The resistive index in renal Doppler sonography: where do we stand? AJR Am J Roentgenol. 2003 Apr;180(4):885-92. doi: 10.2214/ajr.180.4.1800885. No abstract available. PMID 12646425
- [Result] Tang SC, Chan GC, Lai KN. Recent advances in managing and understanding diabetic nephropathy. F1000Res. 2016 May 31;5:F1000 Faculty Rev-1044. doi: 10.12688/f1000research.7693.1. eCollection 2016. PMID 27303648
- [Result] Mancini M, Masulli M, Liuzzi R, Mainenti PP, Ragucci M, Maurea S, Riccardi G, Vaccaro O. Renal duplex sonographic evaluation of type 2 diabetic patients. J Ultrasound Med. 2013 Jun;32(6):1033-40. doi: 10.7863/ultra.32.6.1033. PMID 23716525